CLINICAL TRIAL: NCT03255772
Title: Magnetocardiography Using a Novel Analysis System (Cardioflux) in the Evaluation of Emergency Department Observation Unit Chest Pain Patients
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Collaborators: St. John Hospital & Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1053362-5
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Magnetocardiography; Chest pain
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Chest Pain | interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Acute Chest pain: All patients admitted to the Clinical Decision Unit presenting to the Emergency Department (ED) with chest pain with risk factors suggesting a possible cardiac etiology.
  Interventions: Diagnostic Test: Magnetocardiography

INTERVENTIONS:
Diagnostic Test: Magnetocardiography — Study subjects will be placed within a magnetic shielding apparatus. Noninvasive sensors placed over the subject's torso will acquire magnetic field fluctuations generated by cardiac activity, which will then be analyzed for evidence of myocardial ischemia.
  Other Names: Cardioflux Scan

SUMMARY:
Genetesis is a cardiac diagnostics company which presents a novel magnetocardiogram (MCG) analysis system called CardioFlux. This investigation presents a new, noninvasive diagnostic option to use MCG for rapid diagnosis of acute coronary syndrome. Data from the Cardioflux system will be compared with stress testing methods as well as the results of cardiac catheterization to identify patients with myocardial ischemia.

This is a prospective observational single-blinded convenience pilot study of 100 patients placed in the Clinical Decision Unit (CDU) for evaluation of chest pain at St. John Hospital and Medical Center (Detroit, MI).

Patients enrolled in the study will also have a 30 and 180 day follow up for analysis of adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria: Low and intermediate risk ED patients presenting with chest pain of possible cardiac origin who have a negative first troponin result and non-diagnostic ECG that are to be placed in the Cardiac Diagnostic Unit (CDU) for further evaluation.

Exclusion Criteria:

1. ≤ 18 years of age
2. Patients unable to fit into device
3. Non-ambulatory patients
4. Patients with any implantable device or metal in the thorax area (e.g. pacemaker, AICD, bullet fragments in thorax)
5. Patients with claustrophobia
6. Pregnant women
7. Poor candidate for follow-up
8. Prisoners
9. Repeat participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a pilot study of 100 patients over the age of 18 years who are to be placed in the CDU for evaluation of chest pain of possible cardiac origin will be eligible for the MCG-CF scan based on eligibility criteria criteria.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Identification of Active Myocardial Ischemia | 2 days
  Comparison of Magnetocardiography (MCG) and imaging of myocardial magnetic field/current will be performed directly with standard stress testing protocols performed on patients admitted to a cardiac observation unit.
Identification of Active Myocardial Ischemia | 1 week
  Comparison of Magnetocardiography (MCG) and imaging of magnetic field/current will be directly compared to cardiac catheterization data in those patients who undergo this procedure.

SECONDARY OUTCOMES:
Medium term Adverse Cardiac Events | 6 months
  In patients discharged from the cardiac observation unit with a negative stress test result, how does MCG results correlate with major adverse cardiac events (MACE) at 30 days and 6 months following discharge? MACE will be defined as acute myocardial infarction, coronary revascularization, and all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- St. John Hospital and Medical Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
All patient data will be redacted in terms of name, date of birth and identifying medical record numbers. Patients with specific clinical characteristics may be shared with other researchers if the current protocol is expanded to additional sites or continued within the same research site.

REFERENCES:
- [Background] Chen Y, Fan Y, Yin Z, Zhang H, Zhang Y, Han Z, Wang C. Coronary computed tomographic angiography for patients with low-to-intermediate risk chest pain: A systematic review and meta-analysis. Oncotarget. 2017 Jan 10;8(2):2096-2103. doi: 10.18632/oncotarget.13782. PMID 27926497
- [Background] Hollander JE. The continuing search to identify the very-low-risk chest pain patient. Acad Emerg Med. 1999 Oct;6(10):979-81. doi: 10.1111/j.1553-2712.1999.tb01177.x. No abstract available. PMID 10530653
- [Background] Amsterdam EA, Kirk JD, Bluemke DA, Diercks D, Farkouh ME, Garvey JL, Kontos MC, McCord J, Miller TD, Morise A, Newby LK, Ruberg FL, Scordo KA, Thompson PD; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Cardiovascular Nursing, and Interdisciplinary Council on Quality of Care and Outcomes Research. Testing of low-risk patients presenting to the emergency department with chest pain: a scientific statement from the American Heart Association. Circulation. 2010 Oct 26;122(17):1756-76. doi: 10.1161/CIR.0b013e3181ec61df. Epub 2010 Jul 26. PMID 20660809
- [Background] Pollack CV Jr, Sites FD, Shofer FS, Sease KL, Hollander JE. Application of the TIMI risk score for unstable angina and non-ST elevation acute coronary syndrome to an unselected emergency department chest pain population. Acad Emerg Med. 2006 Jan;13(1):13-8. doi: 10.1197/j.aem.2005.06.031. Epub 2005 Dec 19. PMID 16365321
- [Background] Brindis RG, Douglas PS, Hendel RC, Peterson ED, Wolk MJ, Allen JM, Patel MR, Raskin IE, Hendel RC, Bateman TM, Cerqueira MD, Gibbons RJ, Gillam LD, Gillespie JA, Hendel RC, Iskandrian AE, Jerome SD, Krumholz HM, Messer JV, Spertus JA, Stowers SA; American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group; American Society of Nuclear Cardiology; American Heart Association. ACCF/ASNC appropriateness criteria for single-photon emission computed tomography myocardial perfusion imaging (SPECT MPI): a report of the American College of Cardiology Foundation Quality Strategic Directions Committee Appropriateness Criteria Working Group and the American Society of Nuclear Cardiology endorsed by the American Heart Association. J Am Coll Cardiol. 2005 Oct 18;46(8):1587-605. doi: 10.1016/j.jacc.2005.08.029. PMID 16226194
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Lim HK, Chung N, Kim K, Ko YG, Kwon H, Lee YH, Kim JB, Cho JR, Kim JM, Kim IS, Park YK. Reproducibility of quantitative estimate of magnetocardiographic ventricular depolarization and repolarization parameters in healthy subjects and patients with coronary artery disease. Ann Biomed Eng. 2007 Jan;35(1):59-68. doi: 10.1007/s10439-006-9210-9. Epub 2006 Nov 7. PMID 17089073
- [Background] Goernig M, Liehr M, Tute C, Schlosser M, Haueisen J, Figulla HR, Leder U. Magnetocardiography based spatiotemporal correlation analysis is superior to conventional ECG analysis for identifying myocardial injury. Ann Biomed Eng. 2009 Jan;37(1):107-11. doi: 10.1007/s10439-008-9598-5. Epub 2008 Nov 18. PMID 19015988
- [Background] Tolstrup K, Madsen BE, Ruiz JA, Greenwood SD, Camacho J, Siegel RJ, Gertzen HC, Park JW, Smars PA. Non-invasive resting magnetocardiographic imaging for the rapid detection of ischemia in subjects presenting with chest pain. Cardiology. 2006;106(4):270-6. doi: 10.1159/000093490. Epub 2006 May 29. PMID 16733351